CLINICAL TRIAL: NCT06895642
Title: Development of an Active Video-Based High-Intensity Interval Exercise System in Children With Asthma and Investigation of Immediate Responses
Brief Title: Development of an Active Video-Based High-Intensity Interval Exercise System in Children With Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Manisa Celal Bayar University (Other)
Responsible Party: Principal Investigator, Melissa Köprülüoğlu, Associate Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IzmirKCU302
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Asthma in Children
Keywords: high intensity interval training; video-based exercise; asthmatic children; immediate response
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised controlled interventional study
Who Masked: Participant
Masking Description: Participants only know that they will perform a treadmill and video-based high-intensity interval exercise. They will randomize as video-based or conventional high-intensity interval exercise groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video-based High Intensity Interval Training (Experimental): Participants in this group will perform a video feedback and treadmill-based exercise.
  Interventions: Other: Exercise
- Conventional High Intensity Interval Training (Active Comparator): Participants in this group will perform a treadmill-based exercise.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — After all of the participants perform a symptom-limited cardiopulmonary exercise test, they included a single session high intensity interval exercise created according to test results. They randomized to two gorups as video and treadmill-based or only treadmill-based high intensity interval exercise.

SUMMARY:
The aim of the study was to develop an active video-based high-intensity interval exercise system for the rehabilitation programs of children with asthma and to compare its immediate effects on heart rate variability, hemodynamic responses and thermal responses with a conventional high-intensity interval exercise.

DETAILED DESCRIPTION:
The research consists of two main stages. For the first stage, an active video-based high-intensity interval exercise system will be developed. The game to be developed is considered as an entertaining supporter that adjusts the exercise intensity with the data by the heart rate sensor, warns with visual cues when the child needs to increase the exercise intensity, and keeps the child engaged in the exercise. The second stage is planned to compare the exercise system with the conventional high-intensity interval exercise method that has the same features.

The patient follow-up process will be monitored as; the patient who meets the inclusion and exclusion criteria will be directed by the physician, the patient and family consent will be obtained, pre-intervention evaluation, randomization, intervention, and post-intervention evaluation. The entire process will be carried out in one day.

The patients will be randomized into two groups: conventional high-intensity interval exercise and game-based high-intensity interval exercise, before the evaluation with the closed envelope method. Exercise will be applied at equal intensity (85% of the maximum heart rate) and duration for both groups, and the heart rate of the game-based group will be monitored with the sensor integrated into the game.

ELIGIBILITY:
Inclusion Criteria:

* Having asthma diagnosis according to GINA criteria
* Being between 8-15 years of age
* Having stabil asthma
* Coming to routine follow-ups regularly
* Being under regular pharmacological treatment and having good compliance with treatment confirmed by a physician
* Volunteering to participate in the study (both child and parent)

Exclusion Criteria:

* Having another diagnosed chronic disease other than asthma
* Obesity (Body mass index over 25
* Not having stable asthma defined as having had an exacerbation in the last 4 weeks
* Having severe persistent asthma
* Having exercise-induced asthma
* Not being able to complete the exercise capacity test
* Not being able to maintain the intensity of exercise ±5%

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | Before exercise immediately (in one minute), after exercise immediately (in one minute), and 5th and 10th minutes of the recovery period
  Heart rate variability will be measured in one minute immediately before exercise, in one minute immediately after exercise, and 5 and 10 minutes during recovery with Polar H10.
Heart rate | Before exercise immediately (in one minute), after exercise immediately (in one minute), and 5th and 10th minutes of the recovery period
  Heart rate will be measured in one minute immediately before exercise, in one minute immediately after exercise, and 5 and 10 minutes during recovery with Polar H10.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No